CLINICAL TRIAL: NCT02469662
Title: Retrospective and Prospective Clinical Outcomes Study of the Zimmer® Nexel™ Total Elbow
Brief Title: Clinical Outcomes Study of the Nexel Total Elbow
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMU2014-06E
Record Dates: First submitted 2015-06-08; First posted 2015-06-11 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Elbow Joint Destruction; Post-traumatic Lesions; Ankylosed Joints; Advanced Rheumatoid Arthritis; Joint Instability or Loss of Motion; Acute Comminuted Articular Fracture of Elbow Joint Surfaces; Bone Loss Contributing to Elbow Instability; Bilateral Ankylosis From Causes Other Than Active Sepsis; Post-traumatic Arthritis; Degenerative Arthritis
Keywords: Total Elbow Arthroplasty; TEA; Elbow Arthroplasty; Elbow Replacement; Advanced Rheumatoid Arthritis; Post-Traumatic Arthritis; Degenerative Arthritis; Elbow Joint Destruction; Post-Traumatic Lesions or Bone Loss; Ankylosed Joints; Acute Comminuted Articular Fracture; Significantly compromises daily living activities; Joint or soft tissue damage; Precludes less radical procedures; 13-C3 fractures of the distal humerus
MeSH Terms: conditions — Ankylosis; Joint Instability; Osteoarthritis; Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Retrospective (Experimental): Patients who have had primary or revision total elbow arthroplasty using the Nexel Total Elbow, and who have surgical details available
  Interventions: Device: Nexel Total Elbow
- Prospective (Experimental): Patients who are having primary or revision total elbow arthroplasty who will receive the Nexel Total Elbow
  Interventions: Device: Nexel Total Elbow

INTERVENTIONS:
Device: Nexel Total Elbow — Nexel Total Elbow used in primary or revision total elbow arthroplasty
  Other Names: Nexel Elbow; Nexel

SUMMARY:
The objectives of the study are to confirm safety and performance of the Zimmer Nexel Total Elbow when used in primary or revision total elbow replacement.

DETAILED DESCRIPTION:
The objectives of the study are to confirm safety and performance of the Zimmer® Nexel™ Total Elbow when used in primary or revision total elbow replacement by analysis of standard scoring systems, radiographs, and adverse event records.

The safety of the device will be monitored using the frequency and incidence of reporting adverse events.

The performance of the device will be evaluated by assessing the pain and functional performance, survival of the device, patient health status, and radiographic success of the implant.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older.
* Patient must have signed Institutional Review Board (IRB)/Ethics Committee (EC)-approved informed consent.
* Patient is a candidate for primary or revision total elbow arthroplasty, based on symptoms including at least one of the following:

  * Elbow joint destruction which significantly compromises daily living activities
  * Post-traumatic lesions or bone loss contributing to elbow instability
  * Ankylosed joints, especially cases of bilateral ankylosis from causes other than active sepsis
  * Advanced rheumatoid arthritis, post-traumatic, or degenerative arthritis with incapacitating pain
  * Instability or loss of motion when the degree of joint or soft tissue damage precludes reliable osteosynthesis
  * Acute comminuted articular fracture of elbow joint surfaces that precludes less radical procedures, including 13-C3 fractures of the distal humerus
* Patient is willing and able to complete scheduled follow-up evaluations as defined by the protocol.

Additional Retrospective Arm Inclusion Criteria

* Patient must have undergone a total elbow replacement with the Nexel system between July 2013 and the date of the site initiation visit.
* Patient information available for each retrospective patient must, at minimum, include preoperative demographic information, preoperative physical exam information, the index surgery operative report, and details of the devices implanted.

Exclusion Criteria:

* Patient has a currently active or history of repeated local infection at the surgical site.
* Patient has a current major infection distant from the operative site.
* Patient has a history of prior sepsis.
* Patient suffers from paralysis or dysfunctional neuropathy at the elbow joint.
* Patient has significant ipsilateral hand dysfunction.
* Patient has excessive scarring near the surgical site, which could prevent adequate soft tissue coverage.
* Patient participates in daily activities that may cause significant stress to an implanted device such as heavy labor, torsional stress, and/or competitive sports.
* Patient is a prisoner.
* Patient is mentally incompetent or unable to understand what participation in the study entails.
* Patient is a known alcohol or drug abuser.
* Patient is anticipated to be non-compliant.
* Patient is known to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 10 years
  Based on removal or intended removal of the device and determined using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, MS, Study Director — Zimmer Biomet
Locations (11):
- United States (4):
  - Panorama Orthopedics and Spine Center, Golden, Colorado
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Rothman Institute, Philadelphia, Pennsylvania
  - Campbell Clinic, Germantown, Tennessee
- Sydney Shoulder & Elbow, NSW, Sydney, New South Wales, Australia
- Coxa Hospital, Tampere, Finland
- Hôpital Purpan (Centre Hospitalier Universitaire Toulouse), Toulouse, France
- Arcus Sportklinik, Pforzheim, Germany
- AO Mauriziano, Torino, Italy
- Amphia Ziekenhuis Breda, Breda, Netherlands
- Wrightington, Wigan, United Kingdom